CLINICAL TRIAL: NCT04655586
Title: Assessing Safety, Hospitalization and Efficacy of rNAPc2 in COVID-19 (ASPEN-COVID-19)
Brief Title: Assessing Safety, Hospitalization and Efficacy of rNAPc2 in COVID-19
Acronym: ASPEN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ARCA Biopharma, Inc. (Industry)
Collaborators: Colorado Prevention Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAPc-201/301
Record Dates: First submitted 2020-12-02; First posted 2020-12-07 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-10

CONDITIONS: Covid19
Keywords: D-dimer; Thromboprophylaxis; Anti-coagulant; Thrombotic Events; Coagulation; Inflammation; Heparin
MeSH Terms: conditions — COVID-19; Thrombosis; Inflammation | interventions — anti-coagulant protein C2, Ancylostoma caninum; Heparin

STUDY DESIGN:
Intervention Model Description: investigational product compared to active comparator
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant, clinical events committee members will be blind to treatment assignment. Investigator assessing outcomes will be blinded wherever possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- rNAPc2 Higher Dose (Experimental): loading dose of 7.5 μg/kg SC on Day 1 followed by 5 μg/kg SC on Days 3 and 5
  Interventions: Drug: rNAPc2
- rNAPc2 Lower Dose (Experimental): loading dose of 5 ug/kg SC on Day 1 followed by 3 ug/kg SC on Days 3 and 5
  Interventions: Drug: rNAPc2
- Heparin (Active Comparator): heparin at either prophylactic or therapeutic doses per Standard of Care at Institution
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: rNAPc2 — two dose levels of rNAPc2
  Other Names: AB201; Recombinant Nematode Anticoagulant Protein c2
  Arms: rNAPc2 Higher Dose; rNAPc2 Lower Dose
Drug: Heparin — standard of care heparin per institution (therapeutic or prophylactic regimen)
  Arms: Heparin

SUMMARY:
Sequential randomized, multicenter, active comparator study to evaluate the hypothesis that rNAPc2 (AB201), a novel, potent and highly selective tissue factor inhibitor with anticoagulant, anti-inflammatory and potential antiviral properties, shortens time to recovery compared to heparin in hospitalized patients with COVID-19 and elevated D-dimer levels.

DETAILED DESCRIPTION:
Sequential randomized, multicenter, active comparator study to evaluate the hypothesis that rNAPc2, a novel, potent and highly selective tissue factor inhibitor with anticoagulant, anti-inflammatory and potential antiviral properties, shortens time to recovery compared to heparin in hospitalized patients with COVID-19 and elevated D-dimer levels. Study participants and Clinical Endpoint Committee (CEC) members assessing the clinical endpoints will be blinded to treatment assignment. The protocol comprises sequential Phase 2b and Phase 3 studies. Analysis of Phase 2b data could lead to study discontinuation, adjustment of eligibility criteria or sample size, and will inform the rNAPc2 dose level to be studied in Phase 3.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 90 years at the Screening assessment
2. Weight ≥ 50 kg at randomization
3. Hospitalized with a diagnosis of COVID-19 and in need of inpatient medical care
4. Positive for SARS-CoV-2 on nasopharyngeal, oropharyngeal or other tissue/body fluid samples by PCR or validated other test of ongoing infection (not an antibody test for prior exposure), within seven (7) days of hospitalization or screening assessment
5. D-dimer level > upper limit of normal at screening
6. Provided electronic or written informed consent, either personally or through a legally authorized representative (LAR)
7. Must agree not to participate in a concurrent interventional study involving anticoagulation or anti-platelet therapy
8. Female patients of reproductive or child-bearing potential must be willing to use an effective method of contraception for the duration of the study, and male patients must be willing to use an effective method of contraception to avoid partner pregnancy and abstain from sperm donation for at least 90 days after last dose

Exclusion Criteria:

1. High bleeding risk, e.g. major surgery within prior 1 month, history of a major bleed while receiving anticoagulation, recent hemorrhagic stroke, current or planned (during current hospitalization) dual anti-platelet therapy, platelet count <25,000/uL, current therapeutic anticoagulation for a medical indication other than COVID-19, e.g. atrial fibrillation, known thrombosis, hereditary or acquired coagulopathy treated with therapeutic anticoagulation. Patients receiving prophylactic anticoagulation are eligible if they are willing to discontinue current anticoagulation.
2. Sustained systolic blood pressure < 90 mmHg considered to be clinically significant
3. Persistent eGFR <20 ml/min/1.73m2
4. Known severe liver disease (e.g. bilirubin >3.5 mg/dL (60 umol/L))
5. Life expectancy estimated to be < 72 hours based on current clinical condition
6. Anticipated hospital discharge or transfer within 5 days based on current clinical condition
7. Known anti-phospholipid syndrome
8. Unable to receive heparin, e.g. history of heparin-induced thrombocytopenia and thrombosis (HITT)
9. Participation in any interventional clinical study with an investigational product within seven (7) days of the Screening assessment or within 5 half-lives of the investigational agent, whichever is longer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2022-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bonaca, MD, MPH, Principal Investigator — CPC Clinical Research
Locations (24):
- United States (11):
  - ARCA Investigational Site #119, Fairhope, Alabama
  - ARCA Investigational Site #118, Phoenix, Arizona
  - ARCA Investigational Site #120, Tucson, Arizona
  - ARCA Investigational Site #104, Aurora, Colorado
  - ARCA Investigational Site #117, Denver, Colorado
  - ARCA Investigational Site #101, Jacksonville, Florida
  - ARCA Investigational Site #128, Evanston, Illinois
  - ARCA Investigational Site #113, New Orleans, Louisiana
  - ARCA Investigational Site #105, Falls Church, Virginia
  - ARCA Investigational Site #114, Richmond, Virginia
  - ARCA Investigational Site #103, Tacoma, Washington
- Argentina (8):
  - ARCA Investigational Site #127, San Nicolás de los Arroyos, Buenos Aires
  - ARCA Investigational Site #130, Rosario, Santa Fe Province
  - ARCA Investigational Site #112, Rosario, Sante Fe
  - ARCA Investigational Site #111, Buenos Aires
  - ARCA Investigational Site #115, CABA
  - ARCA Investigational Site #126, Córdoba
  - ARCA Investigational Site #106, San Miguel de Tucumán
  - ARCA Investigational Site #129, San Miguel de Tucumán
- Brazil (5):
  - ARCA Investigational Site #125, Campo Grande, Mato Grosso do Sul
  - ARCA Investigational Site #124, Bragança Paulista, São Paulo
  - ARCA Investigational Site #122, São José do Rio Preto, São Paulo
  - ARCA Investigational Site #123, Porto Alegre
  - ARCA Investigational Site #121, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hess CN, Hsia J, Carroll IA, Nehler MR, Ruf W, Morrow DA, Nicolau JC, Berwanger O, Szarek M, Capell WH, Johri S, Pursley MS, Gupta R, Meehan PS, Franchi F, Effron MB, Marshall D, Graybill CA, Huebler SP, Keuer T, Bristow MR, Bonaca MP. Novel Tissue Factor Inhibition for Thromboprophylaxis in COVID-19: Primary Results of the ASPEN-COVID-19 Trial. Arterioscler Thromb Vasc Biol. 2023 Aug;43(8):1572-1582. doi: 10.1161/ATVBAHA.122.318748. Epub 2023 Jun 29. PMID 37381988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were men and women (18 to 90 years) with a confirmed COVID-19 diagnosis requiring inpatient medical care and an elevated D-dimer level at screening. Enrollment began DEC2020 with the last assessment in MAR2022. 160 participants were enrolled at 15 clinical sites in Argentina, Brazil, and the United States. Originally designed as a sequential Phase 2B/3, the Ph2B top line results dictated substantial design changes for progression to Ph3 and the study was concluded at Ph2.
Pre-assignment Details: All study participants provided informed consent for study participation. Eligible participants were randomized (1:1:2) to receive treatment (i.e., rNAPc2 [1 of 2 dose regimens] or heparin). Randomization was centralized and stratified by local laboratory D-dimer level at screening. Study participants and endpoint assessors were blinded to treatment assignment.
Groups:
- rNAPc2 Lower Dose: loading dose of 5 ug/kg SC on Day 1 followed by 3 ug/kg SC on Days 3 and 5
  rNAPc2: two dose regimens of rNAPc2
- rNAPc2 Higher Dose: loading dose of 7.5 μg/kg SC on Day 1 followed by 5 μg/kg SC on Days 3 and 5
  rNAPc2: two dose regimens of rNAPc2
Period: Overall Study
Arm/Group | rNAPc2 Lower Dose | rNAPc2 Higher Dose | Heparin
Started | 40 | 40 | 80
Completed (The primary reason for participants not receiving all three doses of drug and completing the study were hospital discharges.) | 38 | 34 | 75
Not Completed | 2 | 6 | 5
Not completed — Physician Decision | 1 | 3 | 4
Not completed — Withdrawal by Subject | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: The study was designed as a sequential Phase 2B/3 trial whereby both trial phases were nested in a common protocol. When the 2B top line results dictated substantial design changes for progression to Phase 3 the study was concluded as a Phase 2 trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | rNAPc2 Lower Dose | rNAPc2 Higher Dose | Heparin | Total
Number analyzed (Participants) | 40 | 40 | 80 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 53 | 113
  >=65 years | 10 | 10 | 27 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (13.29) | 52.8 (12.6) | 57.6 (12.8) | 55.5 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 32 | 69
  Male | 24 | 19 | 48 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 1 | 4
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 10 | 8 | 16 | 34
  White | 27 | 32 | 62 | 121
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 1 | 1 | 2 | 4
  United States | 38 | 38 | 74 | 150
  Brazil | 1 | 1 | 4 | 6
WHO COVID Severity [Count of Participants; unit: Participants] — WHO COVID Clinical Improvement scale: severe = oxygen flow rate >=20 L/min, CPAP/BiPAP, mechanical ventilator (from Vital Signs eCRF), vasopressors (dopamine, epinephrine, norepinephrine, phenylephrine) (from Concomitant Medication eCRF). Mild if none of the criteria.
  Participants
    Mild | 26 | 22 | 50 | 98
    Severe | 14 | 18 | 30 | 62
D-Dimer (ng/mL) [Mean (Standard Deviation); unit: ng/mL] | 450.8 (533.8) | 517.4 (588.3) | 864.2 (1794.8) | 680.1 (1354)
D-dimer stratification (%) [Count of Participants; unit: Participants]
  <= 2x Upper limit of normal | 18 | 20 | 35 | 73
  > 2x Upper limit of normal | 22 | 20 | 45 | 87
ACTT Scale [Count of Participants; unit: Participants] — ACTT: adaptive COVID-19 Treatment Trial Score: ACTT scale: 1 = Death, 2 = Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation, 3 = Hospitalized, on non-invasive ventilation or high flow oxygen devices, 4 = Hospitalized, requiring supplemental oxygen, 5 = Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care , 6 = Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care, 7 = Not hospitalized, limitation on activities and/or requiring home oxygen, 8 = Not hospitalized, no limitations on activities.
  Participants
    1 | 0 | 0 | 0 | 0
    2 | 0 | 0 | 2 | 2
    3 | 6 | 5 | 12 | 23
    4 | 10 | 10 | 13 | 33
    5 | 1 | 1 | 3 | 5
    6 | 0 | 0 | 0 | 0
    7 | 0 | 0 | 1 | 1
    8 | 0 | 0 | 0 | 0
    Missing | 23 | 24 | 49 | 96

OUTCOME MEASURES:

1. Primary Outcome: Proportional Change in D-dimer Level From Baseline to Day 8, or Day of Discharge if Prior to Day 8 (Phase 2b)
Description: Proportional change is represented as percent change, and is defined as: 100 × (D-Dimer level at Day 8 or early discharge - D-Dimer level at baseline) / D-Dimer level at baseline. Baseline and post-baseline D-Dimer results are tested in the same laboratory, i.e. both from central laboratory, or local laboratory paired samples if the central laboratory values are not available.
Time Frame: 8 days
Population: Participants included in analysis for whom paired lab results were available.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | rNAPc2 Lower Dose | rNAPc2 Higher Dose | Heparin
Number analyzed (Participants) | 33 | 32 | 70
Percent change | 137 (422.3) | 41.4 (194.6) | 34.7 (133.2)
Statistical Analysis 1: Comparison: rNAPc2 Lower Dose vs rNAPc2 Higher Dose vs Heparin; All rNAPc2 doses (lower and higher) were pooled and compared to Heparin for statistical analysis presentation; Test type: Superiority; p = 0.4715, Wilcoxon Rank Sum — All rNAPc2 vs. Heparin

2. Secondary Outcome: Proportional Change in D-dimer Level From Baseline to 24 Hours Post-dose (Day 2) and Day 3 (Phase 2b)
Description: Proportional change is represented as percent change, and is defined as: 100 × (D-Dimer level at Day 2/3 or early discharge - D-Dimer level at baseline)/D-Dimer level at baseline. Baseline and post-baseline D-Dimer results are tested in the same laboratory.
Time Frame: 2 days and 3 days
Population: Participants included in analysis for whom paired lab results were available.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | rNAPc2 Lower Dose | rNAPc2 Higher Dose | Heparin
Number analyzed (Participants) | 29 | 23 | 55
percentage change
  Day 2 (24h post D1 dose): number analyzed (Participants) | 23 | 23 | 42
  Day 2 (24h post D1 dose) | 23.9 (213.9) | -0.1 (40.3) | 43.5 (317.5)
  Day 3 (48h post D1 dose) | 65.8 (264.5) | -2.3 (68.5) | 21.5 (147.3)
Statistical Analysis 1: Comparison: rNAPc2 Lower Dose vs rNAPc2 Higher Dose vs Heparin; All rNAPc2 doses (lower and higher) were pooled and compared to Heparin for statistical analysis presentation; Test type: Superiority; p = 0.1883, Wilcoxon Rank Sum

3. Secondary Outcome: Number of Major or Non-major Clinically Relevant Bleeding Events Within Eight (8) Days of Randomization as Compared to Heparin (Phase 2b)
Description: Clinical events as reported by site. ISTH= International Society on Thrombosis and Haemostasis, TIMI= Thrombolysis in Myocardial Infarction. Heparin Dosing Strategy as indicated by Investigator. Where subjects have more than one bleeding event recorded, only the highest level of severity was summarized.
Time Frame: 8 days
Population: Safety population includes all participants who were randomized and received at least one dose or part of a dose of study treatment post-randomization. Participants were analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | rNAPc2 Lower Dose | rNAPc2 Higher Dose | Heparin
Number analyzed (Participants) | 38 | 38 | 80
Participants
  ISTH Major or Non-Major Clinically Relevant | 0 | 0 | 1
  Subjects with any ISTH if Major | 1 | 0 | 1
  TIMI Major | 0 | 0 | 1
  TIMI Minor | 0 | 0 | 0
  TIMI Medical attention | 0 | 0 | 0
  TIMI Minimal | 1 | 0 | 0

4. Secondary Outcome: Number of Major or Non-major Clinically Relevant Bleeding Events With rNAPc2 vs. Heparin Through Day 30 (Phase 2b)
Description: as for outcome 3
Time Frame: 30 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | rNAPc2 Lower Dose | rNAPc2 Higher Dose | Heparin
Number analyzed (Participants) | 38 | 38 | 80
Participants
  ISTH Major or Non-Major Clinically Relevant | 1 | 1 | 1
  ISTH Major | 0 | 1 | 1
  ISTH Non-major Clinically Relevant | 1 | 0 | 0
  ISTH Not Clinically Relevant | 2 | 1 | 0
  Subjects With Any ISTH if Major | 3 | 2 | 1
  TIMI Major | 0 | 0 | 1
  TIMI Minor | 0 | 1 | 0
  TIMI medical attention | 1 | 0 | 0
  TIMI Minimal | 2 | 1 | 0

5. Secondary Outcome: Change in High Sensitivity C-reactive Protein Laboratory Values From Baseline Through Day 8 (Phase 2b)
Description: Central lab samples collected per protocol. Proportional change is represented as percent change, and is defined as: 100 × (Biomarker level at Day 8 or early discharge - Biomarker level at baseline)/Biomarker level at baseline.
Time Frame: 8 days
Population: Results analyzed from participants with available lab results.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | rNAPc2 Lower Dose | rNAPc2 Higher Dose | Heparin
Number analyzed (Participants) | 26 | 25 | 50
percent change | -26.1 (203.9) | 270.9 (1556.8) | 12.8 (226.3)
Statistical Analysis 1: Comparison: rNAPc2 Lower Dose vs rNAPc2 Higher Dose vs Heparin; All rNAPc2 doses (lower and higher) were pooled and compared to Heparin for statistical analysis presentation; Test type: Superiority; p = 1.0, Wilcoxon Rank Sum

6. Secondary Outcome: Change in Interleukin-6 Laboratory Values From Baseline Through Day 8 (Phase 2b)
Description: as for outcome 5
Time Frame: 8 days
Population: Results analyzed from participants with available lab results.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | rNAPc2 Lower Dose | rNAPc2 Higher Dose | Heparin
Number analyzed (Participants) | 15 | 17 | 32
percentage change | 317.4 (821.7) | 768.1 (1798.3) | 8.4 (113.8)
Statistical Analysis 1: Comparison: rNAPc2 Lower Dose vs rNAPc2 Higher Dose vs Heparin; All rNAPc2 doses (lower and higher) were pooled and compared to Heparin for statistical analysis presentation; Test type: Superiority; p = 0.0254, Wilcoxon Rank Sum

7. Secondary Outcome: Change in Tissue Factor Laboratory Values From Baseline Through Day 8 (Phase 2b)
Description: as for outcome 5
Time Frame: 8 days
Population: Results analyzed from participants with available lab results.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | rNAPc2 Lower Dose | rNAPc2 Higher Dose | Heparin
Number analyzed (Participants) | 28 | 26 | 52
percentage change | -21.2 (56.3) | -1.8 (89.2) | 23.3 (103.6)
Statistical Analysis 1: Comparison: rNAPc2 Lower Dose vs rNAPc2 Higher Dose vs Heparin; All rNAPc2 doses (lower and higher) were pooled and compared to Heparin for statistical analysis presentation; Test type: Superiority; p = 0.0535, Wilcoxon Rank Sum

8. Secondary Outcome: Change in Antiphospholipid Antibodies Laboratory Values From Baseline Through Day 8 (Anti-Beta 2 Glycoprotein IgG) (Phase 2b)
Description: Proportional change is represented as percent change, and is defined as: 100 × (Biomarker level at Day 8 or early discharge - Biomarker level at baseline)/Biomarker level at baseline.
Time Frame: 8 days
Population: Results analyzed from participants with available lab results.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | rNAPc2 Lower Dose | rNAPc2 Higher Dose | Heparin
Number analyzed (Participants) | 22 | 17 | 33
percentage change | -24.04 (51.84) | -274.3 (1562.57) | 62.99 (479.75)
Statistical Analysis 1: Comparison: rNAPc2 Lower Dose vs rNAPc2 Higher Dose vs Heparin; All rNAPc2 doses (lower and higher) were pooled and compared to Heparin for statistical analysis presentation; Test type: Superiority; p = 0.8300, Wilcoxon Rank Sum

ADVERSE EVENTS:
Time Frame: All AEs were collected from the time of randomization until the participant completed Day 30 or final contact, whichever was longer. All SAEs were collected from the time of consent until the participant completed Day 30 or final contact, whichever was longer. For most participants the final visit/contact was at Day 30 (up to 40 days after screening) or later if delayed due to challenges reaching the participant or obtaining final follow-up information (up to Day 251).
Description: Participant counts were summarized using frequencies and percentages. A participant was counted only once per category of summarization (e.g., the participant was only counted once in the overall 'Any AE' row and was counted once in each row for the specific AE category reported), and reflected the highest level of severity/relatedness reported. Data includes all participants who were randomized and received at least one dose or part of a dose of study treatment post-randomization.
Arm/Group | rNAPc2 Lower Dose | rNAPc2 Higher Dose | Heparin
All-Cause Mortality (participants affected / at risk) | 5/38 | 5/38 | 6/80
Serious Adverse Events (participants affected / at risk) | 18/38 | 29/38 | 26/80
Other Adverse Events (participants affected / at risk) | 18/38 | 18/38 | 36/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rNAPc2 Lower Dose (N=38) | rNAPc2 Higher Dose (N=38) | Heparin (N=80)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney failure (Renal and urinary disorders) | 3 (3) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 6 (6) | 5 (5)
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Abscess on limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Medical device thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lower extremity edema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Cholecycstitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated transaminase (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic hepatits (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Elevated troponin (Investigations) | 1 (1) | 0 (0) | 0 (0)
Worsening of elevated blood glucose (Investigations) | 0 (0) | 1 (1) | 0 (0)
Atrial fibriallation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Type I diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypovolemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Severe coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rNAPc2 Lower Dose (N=38) | rNAPc2 Higher Dose (N=38) | Heparin (N=80)
COVID-19 Pneumonia (Infections and infestations) | 5 (5) | 4 (4) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 5 (5) | 6 (6)
Metabolism and nutrition disorder (Metabolism and nutrition disorders) | 2 (2) | 8 (8) | 10 (10)
Transaminases increase (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Acute kidney injry (Renal and urinary disorders) | 3 (3) | 5 (5) | 2 (2)
Cardiac disorders (Cardiac disorders) | 1 (1) | 1 (1) | 7 (7)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
General disorders and administrative site conditions (General disorders) | 1 (1) | 3 (3) | 3 (3)
Vascular disorders (Vascular disorders) | 1 (1) | 1 (1) | 5 (5)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT04655586/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT04655586/SAP_001.pdf
  • Informed Consent Form (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT04655586/ICF_002.pdf